CLINICAL TRIAL: NCT03766932
Title: Department of Pulmonary & Critical Care Medicine, Chinese PLA General Hospital
Brief Title: Antigenic and Antibody Detection of Candida
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, wang kaifei, xie lixin, Chinese PLA General Hospital
Other Study IDs: Rapid diagnosis
Record Dates: First submitted 2018-12-05; First posted 2018-12-06 (Actual); Last update posted 2018-12-06 (Actual); Status verified 2018-12

CONDITIONS: To Evaluate the Diagnostic Value of Candida Antigen Antibody Detection for Candida Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Blood culture candida positive group
- Tracheal aspiration candida culture positive group
- Urine candida culture positive group
- Other aseptic humoral candida positive group

SUMMARY:
In this study, a multicenter, prospective, synchronous blind, and controlled study was adopted to set the cut-off values of candida specific IgG, IgM, and Mn with the blood culture results as the gold standard, so as to evaluate the diagnostic value of candida specific IgG, IgM, and Mn levels in candida infection.

1. the cut-off values of serum specific IgG, IgM and Mn of candida sinensis infected population in China were established by comparing the positive results of blood culture of 300 healthy people and 100 patients with positive candida sinensis blood culture as the gold standard and using ROC curve (ROC curve).
2. 100 patients with positive tracheal aspiration culture and 100 patients with positive urine culture were enrolled. Serum levels of candida specific IgG, IgM and Mn were detected, and sensitivity, specificity, positive predictive value, negative predictive value and likelihood ratio of candida specific IgG, IgM and Mn in tracheal aspiration and urine were evaluated.
3. 200 high risk patients with candida infection were enrolled, and the aseptic fluid culture and the simultaneous detection of serum specific IgG, IgM and Mn were adopted to explore the diagnostic value of the detection method.
4. positive candida culture in sputum and positive candida culture in tracheal aspirate were taken as the control group to compare the levels of IgG, IgM and Mn in serum of the two groups, and to explore the diagnostic value of different sampling methods for candida pulmonary infection.

ELIGIBILITY:
Inclusion Criteria:Age: (1) 18-85 years old; (2) Candida positive in aseptic humoral culture

-

Exclusion Criteria:(1) no informed consent has been signed; (2) patients with severe immune deficiency -

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with positive aseptic humoral culture among hospitalized patients.The control group were volunteers for outpatient or physical examination
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Serum specific IgG, IgM and Mn levels in the enrolled population | 1-2 years
  ELISA was used to detect the samples

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Pulmonary and Critical Care Medicine, Chinese PLA General Hospital, Beijing, Beijing Municipality, China